CLINICAL TRIAL: NCT04750980
Title: Microbiota as Potential Target for Innovative Preventive and Therapeutic Strategies for Food Allergy
Brief Title: Microbiota and Allergy
Acronym: MATFA I
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, Associate Professor, Federico II University
Other Study IDs: 02e14
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Food allergy: Childen with food allergy
  Interventions: Other: food allergy
- Respiratory allergy: Children with respiratory allergy
  Interventions: Other: respiratory allergy
- Healthy controls: Healthy subjects
  Interventions: Other: healthy controls

INTERVENTIONS:
Other: food allergy — food allergy
  Groups: Food allergy
Other: respiratory allergy — respiratory allergy
  Groups: Respiratory allergy
Other: healthy controls — healthy controls
  Groups: Healthy controls

SUMMARY:
Food allergy derives from a dysregulation of oral tolerance mechanisms. Studies suggest a crucial role for gut microbiota in oral tolerance development. An altered composition of gut microbiota results in an unbalanced local and systemic immune response to food allergens. There are qualitative and quantitative differences in gut microbiota composition in children with food allergy. Preliminary results of MATFA study demonstrated gut microbiota in allergic children.These findings support the pivotal role of the gut microbiota in the pathogenesis of allergic diseases and may open new strategies in the development of innovative preventive and therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Children with sure diagnosis of food allergy,
* children with sure diagnosis of respiratory allergy

Exclusion Criteria:

* age at enrollment <48 months or >84 months;
* eosinophilic disorders of the gastrointestinal tract;
* chronic systemic diseases;
* congenital cardiac defects;
* acute or chronic infections;
* autoimmune diseases;
* immunodeficiencies;
* chronic inflammatory bowel diseases;
* celiac disease;
* cystic fibrosis or other forms of primary pancreatic insufficiency;
* genetic and metabolic diseases;
* food intolerances;
* malignancy;
* chronic pulmonary diseases;
* malformations of the respiratory tract or of the gastrointestinal tract;
* pre-, pro- or sinbiotic use in the previous 3 months;
* antibiotics or gastric acidity inhibitors use in the previous 3 months.

Ages: 48 Months to 84 Months | Sex: All
Age Groups: Child
Study Population: Children with food allergy, children with respiratory allergy and health controls aged 48-84 months
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of gut microbiome features in allergic children and in healthy controls. | at enrollment
  Comparatively evaluation of gut microbiome features in allegic children and in healthy controls.

SECONDARY OUTCOMES:
Gut microbiome and allergy disease course | at enrollment
  Evaluation of gut microbiome influence on allergy disease course
Evaluation of gut microbiome features in children affected by different allergies (food and respiratory) | at enrollment
  Comparatively evaluation of gut microbiome features in children with different allergies (food and respiratory)
Evaluation of gut microbiome features in children affected by different type of food allergy | at enrollment
  Evaluation of gut microbiome features in children affected by different type of food allergy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Filippis F, Paparo L, Nocerino R, Della Gatta G, Carucci L, Russo R, Pasolli E, Ercolini D, Berni Canani R. Specific gut microbiome signatures and the associated pro-inflamatory functions are linked to pediatric allergy and acquisition of immune tolerance. Nat Commun. 2021 Oct 13;12(1):5958. doi: 10.1038/s41467-021-26266-z. PMID 34645820